CLINICAL TRIAL: NCT06640348
Title: Ultrasensitive SERS Platform With Highly Efficient Enrichment of Analyte for Screening and Diagnosis of Epithelial Ovarian Cancer
Status: Recruiting | Type: Observational
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: YingZhou 2024-10
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Ovarian Cancer, Epithelial
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy control: By analyzing the Raman signals of peripheral serum from normal controls, unique signal characteristics specific to ovarian cancer patients are identified through comparative analysis with the control group.
  Interventions: Other: No intervention
- Ovarian cancer group: Extract information from blood samples of ovarian cancer patients, specifically identifying cancer and non-cancer signals to construct a statistical algorithm model for the early diagnosis of ovarian cancer.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This project is an open, single-center, prospective study aimed at developing high-sensitivity, high-specificity enrichment SERS chips using femtosecond laser processing technology. It involves extracting information from blood samples of ovarian cancer patients and normal controls, specifically identifying cancer and non-cancer signals. The study will construct a statistical algorithm model for the early diagnosis of ovarian cancer, enabling early identification and intervention for ovarian cancer patients.

DETAILED DESCRIPTION:
Epithelial Ovarian Cancer (EOC) poses a significant challenge in the field of gynecological oncology regarding precise early screening. In response to this critical scientific issue, the research team has designed and developed a high-sensitivity, high-specificity enrichment SERS chip, exploring its applications in the screening and diagnosis of ovarian cancer. The development of the SERS chip and its functional implementation has been done.Clinical research trials are conducted for ovarian cancer screening and diagnosis, analyzing the physicochemical properties of key biomolecules in the blood of ovarian cancer patients. The study reveals the interaction patterns between SERS active particles and biomolecules, establishing a competitive adsorption model between multiple biomolecules and active particles. Raman spectra of individual components are collected to create a characteristic Raman information database for key biomolecules.

The analysis of Raman spectra from ovarian cancer patients and healthy individuals delves into the characteristic signals, constructing a statistical classification model for patient and normal Raman signals. Different tissue types and grades of ovarian cancer patients' Raman spectra signals are analyzed, establishing high-throughput classification methods for various ovarian cancers. By combining clinical gold-standard detection techniques, the sources of characteristic signals are determined, providing a theoretical foundation and technical support for conducting ovarian cancer research and establishing treatment plans in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects understand the trial process, sign the informed consent form, voluntarily participate in the study, and are capable of following the protocol;
2. Aged 18 to 70 (inclusive):

Cancer group: Ovarian cancer patients (50 cases of high-grade serous ovarian cancer, 15 cases of low-grade serous ovarian cancer, 20 cases of endometrioid ovarian cancer, 20 cases of clear cell carcinoma) i. All ovarian cancer patients are initial treatment patients with complete clinical data; ii. Patients have an ECOG performance status score of 0-3 and a life expectancy of more than 6 months; iii. Subjects consent to blood sample collection for SERS analysis (provided free of charge); iv. Good organ function.

Normal control group: (20 cases) i. Normal control subjects are patients undergoing surgery for benign diseases; ii. Patients have complete clinical data; iii. Subjects have not undergone any radical treatment for the benign lesion prior to blood collection.

Exclusion Criteria:

1. Severe or uncontrolled diseases, including but not limited to: uncontrollable nausea and vomiting, gastrointestinal diseases that may interfere with drug absorption and metabolism, mental illnesses affecting the patient's ability to sign the informed consent form, a history of severe cardiovascular disease, infectious diseases (such as syphilis, AIDS, active hepatitis C, or active hepatitis B), infectious conditions (such as abscesses), or active rheumatic diseases, etc.;
2. A history of blood transfusion within 4 weeks prior to the study;
3. Pregnant, postpartum, or breastfeeding patients, or patients planning to become pregnant during the study treatment;
4. Patients with a history of other tumors;
5. The investigator deems the subject unsuitable for participation in this clinical study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects include patients with epithelial ovarian cancer, while the control group consists of patients undergoing surgery for benign diseases.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS PFS | one year
  progression free survival
OS | three year
  OS (overall survival) is defined as the time which begins at diagnosis and up to the time of death

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Provincal Hospital, Hefei, Anhui, China